CLINICAL TRIAL: NCT03380143
Title: Whole-of-Community Systems Intervention for Youth Population Physical Activity
Brief Title: Whole-of-Community Youth Population Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Iowa State University (Other); Kansas State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0446-18-EP
Record Dates: First submitted 2017-12-06; First posted 2017-12-20 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Physical Activity
Keywords: Children; Cancer Prevention; Population Health; Rural; Community; School; After School; Youth Sport; Intervention; Multilevel; Systems
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This design can be described as a staggered-start, stepped-wedge, community randomized trial. The design includes two sequential intervention waves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wellscapes Intervention (Experimental): The wellness landscape intervention (Wellscapes) will establish a multi-level system infrastructure (Community Hub, Organization Wellness Teams, Activity Setting/Leaders) and provide training and support for population health quality improvement cycle processes targeting two evidence-based practices (EBPs): (1) stacking time segments of PA episodes within an organization's daily routine, and (2) improving the quality of PA episodes (% time in PA).
  Interventions: Behavioral: Wellness Landscape Intervention
- Standard Practice (Active Comparator): The standard collective impact public health practice intervention will establish a multi-level system infrastructure and provide training on community development.
  Interventions: Behavioral: Standard Practice

INTERVENTIONS:
Behavioral: Wellness Landscape Intervention — Community and organization systems intervention targeting youth population physical activity
  Other Names: Wellscapes
  Arms: Wellscapes Intervention
Behavioral: Standard Practice — Community development intervention
  Other Names: Collective Impact
  Arms: Standard Practice

SUMMARY:
This study will evaluate the impact of a whole-of-community multi-level adaptive systems intervention on implementation of community change and youth population physical activity. Building on local health department partnerships, the investigators will conduct a two-wave staggered-start community randomized trial with four volunteer rural communities (each having nested school, after-school, scouting/4-H club, youth sport organizations) randomly assigned to intervention or standard public health practice.

DETAILED DESCRIPTION:
The underlying conditions where youth live are associated with population health outcomes, with rural communities facing under-studied challenges. Youth physical activity (PA), a key risk factor linked to later cancer occurrence, is an outcome of community conditions. The proposed work will address a critical public health need by evaluating the impact of a whole-of-community multi-level adaptive systems intervention on implementation of community change and youth population PA. The intervention, Wellscapes, is based on a hierarchical patch dynamics paradigm, given that communities are "wellness landscapes" of spatially heterogeneous geographic areas, characterized by a patchwork of interacting organization and activity settings. The intervention will establish a multi-level system infrastructure (Community Hub, Organization Wellness Teams, Activity Setting/Leaders) and provide training and support for population health quality improvement cycle processes targeting two evidence-based practices (EBPs): (1) stacking time segments of PA episodes within an organization's daily routine, and (2) improving the quality of PA episodes (% time in PA). The omnibus hypothesis is that intervention communities (plus organizations and leaders nested within) will have synergy and capacity to implement EBPs, adapting to continuously changing local system drivers to create a whole-of-community ecosystem of diverse and equitable youth PA opportunities. Building on local health department partnerships, the investigators will conduct a two-wave staggered-start community randomized trial with four volunteer rural communities (each having nested school, after-school, scouting/4-H club, youth sport organizations) randomly assigned to intervention or standard public health practice. For baseline and intervention years, one day per month in the fall (3 days) and spring (3 days), organization activity settings (e.g., classrooms, teams) that house 480 children in 3rd through 6th grades will be assessed, resulting in observed community condition data, PA accelerometer data, and setting reach data (children % attendance by gender, ethnicity, free/reduced lunch status, and grade). The investigators will also obtain estimates of population level PA with the use of the calibrated Youth Activity Profile, as well as community system qualitative data. The specific aims are to: (1) Determine the impact of the intervention on multi-level community system outcomes; and (2) Determine the implementation system drivers of multi-level youth population PA. The investigators will use "big data" multi- level modeling methods for this effectiveness-implementation hybrid design, because there is a dual focus on testing an implementation strategy while simultaneously evaluating youth population PA impact. The research is significant because it evaluates a method for improving population health, theory-based systems, and behavior change processes in low-resource rural communities. The proposed research is novel because the adaptive patch dynamics approach builds capacity for both equitable collaboration and EBPs implementation across multiple local systems that are individually and collectively, dynamic and unpredictable.

ELIGIBILITY:
Inclusion Criteria:

* Community located in rural micropolitan area
* Community is a one high school town
* Organization is a school district
* Organization is a after school program
* Organization is a youth club system
* Organization is a youth sport delivery system
* Leaders of settings in school, after-school, club, and youth sport
* 3rd through 6th grade settings and children within

Exclusion Criteria:

-

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 697 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Change in minutes of moderate-to-vigorous physical activity assessed by accelerometer | Baseline, 12 months
  Average of school class, after-school class, youth club meeting, and youth sport practice physical activity
Change in frequency of implemented episode sessions of physical activity assessed by observation | Baseline, 12 months
  Average of observed frequency of implemented physical activity episodes in school class, after-school class, youth club meeting, and youth sport practices

SECONDARY OUTCOMES:
Change in minutes of moderate-to-vigorous physical activity assessed by self-report | Baseline, 12 months
  Youth Physical Activity Profile

CONTACTS AND LOCATIONS:
Overall Officials: David A Dzewaltowski, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available within 1 year of study completion.
Access Criteria: Data access will be reviewed by investigator team. Requesters will be required to sign data access agreement.

REFERENCES:
- [Background] Kellstedt DK, Schenkelberg MA, Essay AM, Welk GJ, Rosenkranz RR, Idoate R, Ramos AK, Grimm B, Dzewaltowski DA. Rural community systems: Youth physical activity promotion through community collaboration. Prev Med Rep. 2021 Jul 6;23:101486. doi: 10.1016/j.pmedr.2021.101486. eCollection 2021 Sep. PMID 34458077
- [Background] Kellstedt DK, Schenkelberg MA, Essay AM, Von Seggern MJ, Rosenkranz RR, Welk GJ, High R, Dzewaltowski DA. Youth sport participation and physical activity in rural communities. Arch Public Health. 2021 Apr 8;79(1):46. doi: 10.1186/s13690-021-00570-y. PMID 33832548
- [Background] Schenkelberg MA, Essay AM, Rosen MS, Bavari AE, Norgelas SJ, Rosenkranz RR, Welk GJ, Dzewaltowski DA. A protocol for coordinating rural community stakeholders to implement whole-of-community youth physical activity surveillance through school systems. Prev Med Rep. 2021 Aug 26;24:101536. doi: 10.1016/j.pmedr.2021.101536. eCollection 2021 Dec. PMID 34976611
- [Background] Essay AM, Schenkelberg MA, Von Seggern MJ, Rosen MS, Schlechter CR, Rosenkranz RR, Dzewaltowski DA. A Protocol for a Local Community Monitoring and Feedback System for Physical Activity in Organized Group Settings for Children. J Phys Act Health. 2023 Mar 25;20(5):385-393. doi: 10.1123/jpah.2022-0486. Print 2023 May 1. PMID 36965493
- [Background] Kellstedt DK, Essay AM, Schenkelberg MA, Rosen MS, Von Seggern MJ, Idoate R, Welk GJ, Rosenkranz RR, Dzewaltowski DA. COVID-19 pandemic and changes in children's physical activity in a rural US community: a mixed methods study. BMJ Open. 2022 Oct 27;12(10):e062987. doi: 10.1136/bmjopen-2022-062987. PMID 36302579
- [Derived] Rogers AE, Wichman CS, Schenkelberg MA, Dzewaltowski DA. Inequality in Children's Physical Activity Across Time-Segmented Youth Sport Practice. Res Q Exerc Sport. 2025 Mar;96(1):96-108. doi: 10.1080/02701367.2024.2367565. Epub 2024 Jul 11. PMID 38990545
- [Derived] Von Seggern MJ, Rogers AE, Schenkelberg MA, Kellstedt DK, Welk GJ, High R, Dzewaltowski DA. Sociodemographic influences on youth sport participation and physical activity among children living within concentrated Hispanic/Latino rural communities. Front Public Health. 2024 Feb 21;12:1345635. doi: 10.3389/fpubh.2024.1345635. eCollection 2024. PMID 38450148